CLINICAL TRIAL: NCT07109609
Title: Topical Menthol for Tear Secretion
Acronym: TMTS
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Reinhold Vieth (Industry)
Collaborators: Stearacl Inc (Industry)
Responsible Party: Sponsor-Investigator, Reinhold Vieth, CEO Stearacl Inc, Canada, Stearacl Inc
Organization: Stearacl Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: M240706
Record Dates: First submitted 2025-07-30; First posted 2025-08-07 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-07

CONDITIONS: Healthy; Dry Eyes
Keywords: tear secretion; dry eyes; eye drops; menthol; vapor; cornea
MeSH Terms: conditions — Dry Eye Syndromes; Corneal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Topical Menthol in Oil (Experimental): Menthol solution rolled onto the cheek below rim of a pair of glasses
  Interventions: Drug: Topical application of 20% menthol solution in MCT oil.
- Topical Placebo Oil only (Placebo Comparator): Oil vehicle only rolled onto the cheek below rim of a pair of glasses
  Interventions: Drug: Topical Placebo Oil rolled onto the cheek.

INTERVENTIONS:
Drug: Topical application of 20% menthol solution in MCT oil. — To facilitate reproducible and correct application of the solution, the subject wears glasses while the product is applied. The solution is rolled onto one cheek by rolling it to an area of about 2cm X 2cm at the cheekbone, underneath the bottom rim of the glasses worn. This method delivers about 12 mg solution, i.e. 2.4 mg menthol to one cheek. Or this method delviers 12 mg of placebo oil. The subject then sits in still air for 5 minutes, at which point tissue is wiped across the skin below the bottom eyelashes to permit the weighing of secreted tear.
  Arms: Topical Menthol in Oil
Drug: Topical Placebo Oil rolled onto the cheek. — To facilitate reproducible and correct application of the Placebo oil, the subject wears glasses while the product is applied. The Placebo oil is rolled onto one cheek by rolling it to an area of about 2cm X 2cm at the cheekbone, underneath the bottom rim of the glasses worn. This method delivers zero active agent. The subject then sits in still air for 5 minutes, at which point tissue is wiped across the skin below the bottom eyelashes to permit the weighing of secreted tear.
  Arms: Topical Placebo Oil only

SUMMARY:
Tears are the natural way to keep eyes moist, and tears are important for good vision and healthy eyes. Eyes without enought tears get dry and sore.

The natural and normal way to stimulate secretion of tears is by turning on cold sensors that are located on the cornea of the eye. Tear are normally released across the eyeball in a finely balanced system that balances out that natural evaporation. But sometimes there is not enough tear secretion to balance out the evaporation of tears and eyes can get sore.

The aim here is to test whether menthol in its vapor form may possibly turn on those cold sensors and thus cause secretion of tears. Use of menthol vapors may be like having a switch to release more tears.

The aim of this clinical trial is to test the hypothesis that a menthol solution applied onto a cheek will release enough menthol vapor into the air flowing up over the eye's cornea to stimulate cold sensors enough to make a tear flow from the eye.

If the hypothesis that menthol safely stimulates tear secretion in healthy people proves to be correct, then this clinical trial may inspire more new research into the use of menthol as an alternative to the use of eye drops for some people.

DETAILED DESCRIPTION:
This is a proof-of-principle clinical trial. It is a double-blind, placebo-controlled, randomized clinical trial. Participants are not being seen by a physician for eye disease, and there is a 50% probability that a participant will receive active treatment, or 50% probability that they will just receive the carrier oil with nothing in it (placebo).

ELIGIBILITY:
Inclusion Criteria:

* Not under care of an opthalmologist for treatment of dry-eyes

Exclusion Criteria:

* • Excluded if "Yes" to any of the questions below.

  * Are you allergic to menthol or to menthol-containing products like tooth paste or certain cold remedies?
  * Are you wearing contact lenses during the time of testing? ________
  * Are there tears present prior to applying the menthol? ________
  * Did you use of eye drops during the hour before participation? ________
  * Do you have broken, irritated, sensitive skin and/or acne at or around application site? ________
  * Do you have a history of atopy, allergic diseases at the skin of your cheeks?
  * Do you have Stevens-Johnson syndrome, which is any known skin response to chemical, thermal, or radiation injury to the application area? ____

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-17 (Actual); Primary Completion 2025-11-07 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective measure of tear stimulation Yes or No | Participant is observed for 5 minutes after application, to record tear-weight data, and the related questions that are asked are completed within 10 minutes after applicaiton.
  The outcome is the binary yes/no observation of active tear secretion that overflows to the skin below the bottom eyelashes. Subject sits in still air while wearing glasses to ensure correct positioning of the topical application. The solution of menthol or placebo is dispensed from a roller-ball bottle to the right eye only, onto an area about 2cm x 2 cm just below the bottom rim of the glasses; that is, inferior to the pupil, and in line with the bottom of the nose. Within 5 minutes of sitting in still air, If moisture is evident below the bottom eyelashes, glasses are removed and tissue is dabbed, or wiped under bottom eyelash to take up the tear. If that wipe increases the weight of the tissue by at least 6 milligrams, then a "Yes" response is recorded. If after 5 minutes a wipe of tissue across the bottom eyelashes of the right eye does not increase the weight of tissue by at least 6 milligrams, a "No" is recorded to indicate that there was no increase in tear secretion.
Weight of tear | Measured at 5 minutes after dose application.
  The actual measured weight of the tear(s) collected onto the tissue, from below the right eye.
Was there a subjective difference between left and right eyes in terms of sense if moisture | 5 to 10 minutes after application
  Response to the question: " Which eye feels more moist? Left eye more moist or No difference (both same) or ….Right eye more moist"
Weight of nasal secretion blown into tissue. | Within 10 minutes of applying the dose.
  The purpose is to test whether there is evidence of shared innervation of TRPM8 receptors (the menthol-responsive sensors for cold) in cornea and nasal subepithelium. The particpant holds closed the left nostril, while blowing into a tissue from the right nostril. The increase in weight of tissue is measured.

SECONDARY OUTCOMES:
Weight of nasal secretion | 5 to 10 minutes after application
  Subject blows their nose into a tissue, and the increase in tissue weight is recorded.
Discomfortable feeling at the treated eye. | 10 minutes
  At your right eye, was there anything uncomfortable feeling? Nothing mild moderate severe (choose one)
Degree of cooling or pain at the skin where the dose was applied. | 10 minutes
  At the skin of the cheek, where it was rolled on, did you feel (choose one) COOLING OR NOTHING OR PAIN If cooling or pain, how strong was the feeling? (choose one) Nothing mild moderate severe
Did the procedure increase sense of runny nose? | 10 minutes
  Did you feel a runny nose, or nasal secretion during the 5 minutes of waiting? No or Yes And if Yes, at which nostril? Left or Right or Both nostrils

CONTACTS AND LOCATIONS:
Locations (1):
- Stearacl Incorporated., Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
A spreadsheet of anonymized IPD collected throughout the trial may be made upon inquiry with the corresponding author of any peer-reviewed publication ensuing from this work.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 1 month after final publication
Access Criteria: The senior author of any ensuing publication will correspond with suitably qualified investigators, to discuss the type and form of data made available.